CLINICAL TRIAL: NCT06555640
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase II Clinical Study to Evaluate the Efficacy and Safety of Subcutaneous Injection of DR10624 in Subjects With Severe Hypertriglyceridemia
Brief Title: A Phase II Study to Evaluate the Efficacy and Safety of of DR10624 in Subjects With Severe Hypertriglyceridemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang Doer Biologics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DR10624-201
Record Dates: First submitted 2024-07-30; First posted 2024-08-15 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Severe Hypertriglyceridemia
MeSH Terms: conditions — Hypertriglyceridemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Cohort 1: DR10624 injection (Experimental): DR10624 injection administered weekly (QW)
  Interventions: Drug: DR10624 Injection
- Cohort 1: Placebo (Placebo Comparator): Placebo administered weekly (QW)
  Interventions: Drug: Placebo
- Cohort 2: DR10624 injection (Experimental): DR10624 injection administered weekly (QW)
  Interventions: Drug: DR10624 Injection
- Cohort 2: Placebo (Placebo Comparator): Placebo administered weekly (QW)
  Interventions: Drug: Placebo
- Cohort 3: DR10624 injection (Experimental): DR10624 injection administered weekly (QW)
  Interventions: Drug: DR10624 Injection
- Cohort 3: Placebo (Placebo Comparator): Placebo administered weekly (QW)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DR10624 Injection — Drug: DR10624 injection
  Arms: Cohort 1: DR10624 injection; Cohort 2: DR10624 injection; Cohort 3: DR10624 injection
Drug: Placebo — Drug: placebo
  Arms: Cohort 1: Placebo; Cohort 2: Placebo; Cohort 3: Placebo

SUMMARY:
DR10624 is an Fc fusion protein tri-agonist with balanced glucagon-like peptide-1 receptor (GLP-1R)/glucagon receptor (GCGR)/ fibroblast growth factor 21 receptor (FGF21R) agonizing activities. The objectives of the planned clinical investigation will be to evaluate the efficacy of DR10624 on fasting serum triglyceride (TG) levels after 12 weeks of treatment in subjects with severe hypertriglyceridemia (SHTG).

DETAILED DESCRIPTION:
The subjects will be randomly assigned to experimental groups and placebo-controlled groups. Each participant will be enrolled in only one cohort.

ELIGIBILITY:
Inclusion Criteria:

* 1.Subjects or their legally acceptable representatives must be able to provide written informed consent, understand the procedures and methods of the study, and agree to comply with all protocol requirements.

  2.Male or female, age of 18 to 75 years (inclusive) at screening.

  3.Subjects must have a BMI of >19 kg/m2 and BMI of ≤45.0 kg/m2 , and body weight ≥50 Kg at screening.

  4.During screening or within 1 week prior to screening, the TG levels should meet the following criteria: 4.80 mmol/L (425 mg/dL) ≤ fasting TG < 22.60 mmol/L (2000 mg/dL).

  5.The average fasting TG level of Visit 2 and Visit 3 values must meet: 5.65 mmol/L (500 mg/dL) ≤fasting TG <22.60 mmol/L(2000 mg/dL); or the average fasting TG level of Visit 3 and Visit 3.1 values must meet the same criteria.

  6.Subjects will able to accept rencommendation on therapeutic lifestyle modificationa and maintain a stable lifestyle for the duration of the study.

  7.Subjects who are receiving statins, cholesterol-absorption inhibitor (CAI), fibrates, niacin ≥500 mg/day, or prescription omega-3 fish oil must have achieved a stable dose for at least 4 weeks before screening.

  8.Subjects diagnosed with type 2 diabetes(T2DM) must have a glycosylated hemoglobin level at screening of<9.5%(80 mmol/mol）and treated with lifestyle modification or a stable doses of antidiabetic medications for at least 8 weeks prior to screening.

Exclusion Criteria:

* 1.Subjects with known familial hyperchylomicronemia (Fredrickson type 1) ,apo c-II deficiency,or familial β-lipoprotein dyslipidemia (Fredrickson type 3); or subjects with a high suspicion of having this three conditions.

  2.Subjects who have lost ≥5% of body weight within 3 months prior to screening, or who lose ≥5% of body weight during screening, or who plan to lose body weight during the study.

  3.Subjects with type 1 diabetes, or nephrotic syndrome.

  4.Subjects with cirrhosis, alcoholic liver disease, liver failure, liver cancer, or autoimmune hepatitis.

  5.Subjects type 2 diabetes with a duration of less than 12 weeks or with severe complications.

  6.Uncontrolled hypertension at screening, defined as systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥100 mmHg under medication conditions.

  7.Subjects with an active or untreated malignancy or who have been in remission from a clinically significant malignancy (other than basal or squamous cell skin cancer, in situ carcinomas of the cervix, or in situ prostate cancer) for <5 years prior to screening.

  8.Subjects with a family or personal history of medullary thyroid carcinoma (MTC),multiple endocrine neoplasia syndrome type 2 (MEN2),severe active or unstable major depressive disorder (MDD), or other serious mental disorders (such as schizophrenia, bipolar disorder, or other severe mood or anxiety disorders) or suicidal.

  9.Subjects with a known clinically significant gastric emptying abnormality (e.g. severe diabetic gastroparesis), and who have undergone or plan to undergo gastric bypass surgery or gastric banding surgery during the study, or those who chronically take drugs that directly affect GI motility.

  10.New York Heart Association Functional Classification III or IV CHF.

  11.In the opinion of the investigator, the subjects are likely to require concurrent treatment with systemic glucocorticoids during the trial due to comorbidities.

  12.Subjects with a history of acute pancreatitis within 1 year prior to screening, or a history of chronic pancreatitis, or symptomatic of gallbladder disease (e.g. choledocholithiasis, gallbladder multiple stones, unless treated with cholecystectomy).

  13.Subjects with any of the following cardiovascular (CV) conditions within 6 months prior to screening: acute myocardial infarction, cerebral hemorrhage or cerebral infarction (except lacunar infarction), or hospitalization due to CHF, unstable angina pectoris or transient ischemic attack, or cardiac surgery such as percutaneous coronary intervention and coronary artery bypass grafting,or subjects who have been treated with GLP-1R agonists, or have participated in a clinical study involving GLP-1R and received the study drug within 6 months prior to screening.

  14.Subjects who have undergone large-sized surgery,have been treated with GCGR or multiple target point and agonists containing FGF-21R targets;have been treated with SiRNA type and monoclonal antibody type of PCSK9 inhibitors;or who have participated in a clinical study related to above all the types of drug within 3 months prior to screening.

  15.Subjects with severe trauma, severe infection who have not recoveredwithin 4 weeks prior to screening,who have been treated with DPP-4 inhibitors, or have participated in a clinical study related to DPP-4 inhibitors and received the study product;who have undergone lipid apheresis or plasma exchange treatment within the last 4 weeks or plan to undergo apheresis or plasma exchange during the study period.

  16.Subjects with hyperthyroidism or hypothyroidism who have the stable dose of therapeutic drugs less than 3 months prior to screening.

  17.Subjects with Cushing's syndrome or who have continuously or cumulatively used systemic glucocorticoids for more than 14 days within 6 months before screening, Inhaled or topical corticosteroids are permitted.

  18.Subjects who do not agree to discontinue medications, supplements, or nutraceuticals that have lipid-altering effects other than those specified in the protocol.

  19.Subjects who are taking insulin or second-generation antipsychotics and cannot stop taking them.

  20.Serum calcitonin ≥20 ng/L (pg/mL) in subjects with eGFR≥60 mL/min/1.73 m2 , or serum calcitonin ≥35 ng/L (pg/mL) in subjects with eGFR <60 mL/min/1.73 m2.

  21.Alanine aminotransferase>3.0 × upper limit of normal value (ULN) and/or aspartate aminotransferase>3.0 × ULN and/or total bilirubin>1.5 × ULN.

  22.Glomerular filtration rate eGFR < 45 mL/min/1.73 m2

  23.TSH > upper normal limit or < lower normal limit.

  24.Serum amylase or lipase > 2.0 × ULN.

  25.Hemoglobin < 110 g/L (males) or < 100 g/L (females).

  26.Test positive for Human Immunodeficiency Virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV), HBV and HCV determined by antibodies first and, if positive, by DNA/ribonucleic acid (RNA).

  27.Clinically significant 12-lead electrocardiogram (ECG) abnormalities at the time of screening.

  28.History of drug abuse or excessive alcohol consumption within 3 months prior to screening.

  29.Presence of potential allergies to the study drug, its ingredients, or drugs of the same class.

  30.Pregnant or lactating women;as well as men and women of childbearing potential who are unwilling to prevent pregnancy throughout the study and within the specified time after the study.

  31.Blood donation and/or blood loss ≥400 mL, or bone marrow donation within 3 months prior to screening.

  32.Subjects in which the investigator deems to that there are any other factors may affect the efficacy or safety evaluation of this study(including medical, psychological, social, or geographical considerations) .

Ages: 17 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-08-29 (Actual)

PRIMARY OUTCOMES:
Change of fasting TG | From baseline to Week 12
  The percentage change of fasting TG in all the participants from baseline to Week 12

SECONDARY OUTCOMES:
Change of lipid profile and lipoprotein profile | From baseline to Week 12
  The percentage change of fasting total cholesterol (TC), low density lipoprotein cholesterol (LDL-C), high density lipoprotein cholesterol (HDL-C), non-high density lipoprotein cholesterol (non-HDL-C), very low density lipoprotein cholesterol (VLDL-C), free fatty acid (FFA), triglyceride rich lipoprotein cholesterol (TRL-C), lipoprotein (a) [Lp(a)], apolipoprotein C3 (Apo C3), apolipoprotein B (Apo B), apolipoprotein B48 (Apo B48), apolipoprotein B100 (Apo B100), apolipoprotein A1 (Apo A1) and apolipoprotein A5 (Apo A5)
Number of participants whose fasting TG lowered by at least 50% | From baseline to Week 12
  The number of participants whose fasting TG decreased by at least 50% from baseline
Change of glycosylated hemoglobin (HbA1C) | From baseline to Week 12
  The change of glycosylated hemoglobin (HbA1C) in all participants
Change of liver fat content | From baseline to week 12
  Measured by magnetic resonance imaging-proton density fat fraction (MRI-PDFF)
Change of liver stiffness measurements (LSM) | From baseline to week 12
  The change of liver stiffness in subjects with baseline hepatic fat fraction of at least 8% measured by FibroScan
Change of controlled decay index (CAP) | From baseline to week 12
  The change of CAP in subjects with baseline hepatic fat fraction of at least 8% measured by MRI-PDFF
Incidence and severity of adverse events | through study completion, up to 17 weeks
  The number of participants with treatment-related adverse events as assessed by CTCAE V5.0, such outcomes are included but not limited to hypoglycemia events, injection site reactions, 12-lead Electrocardiogram (ECG) QTc intervals and vital signs (blood pressure, heart rate, respiratory rate and body temperature), physical examinations and safety laboratory tests, etc.
Anti-drug antibody（ADA） | through study completion, up to 17 weeks
  Anti-drug antibody（ADA）
Pharmacokinetic Ctrough blood concentration of DR10624 | through study completion, up to 17 weeks
  Pharmacokinetic Ctrough blood concentration of DR10624

CONTACTS AND LOCATIONS:
Overall Officials: Jianping Li, M.D., Study Chair — Peking University First Hospital
Locations (35):
- China (35):
  - Baoding No.1 Central Hospital, Baoding
  - The First Affiliated Hospital of Baotou Medical College, Baotou
  - Peking University First Hospital, Beijing
  - The First Affiliated Hospital of Bengbu Medical University, Bengbu
  - The First Hospital of Jilin University, Changchun
  - The Second Hospital of Jilin University, Changchun
  - Second Xiangya Hospital of Central South University, Changsha
  - Chifeng Municipal Hospital, Chifeng
  - Daqing People's Hospital, Daqing
  - The Affiliated Hospital of Hangzhou Normal University, Hangzhou
  - The Fourth Hospital of Harbin Medical University, Harbin
  - The First Affiliated Hospital of South China University, Hengyang
  - Inner Mongolia People's Hospital., Hohhot
  - Huzhou Central Hospital, Huzhou
  - Lishui Municipal Central Hospital, Lishui
  - Luoyang Third Peoples Hospital, Luoyang
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang
  - Meihekou Central Hospital, Meihekou
  - The Second Affiliated Hospital to Nanchang University, Nanchang
  - The Third Hospital of Nanchang, Nanchang
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing
  - The Affiliated Hospital of Nantong University, Nantong
  - Nanyang Central Hospital, Nanyang
  - Panjin Liaoyou Baoshihua Hospital, Panjin
  - Pingxiang People's Hospital, Pingxiang
  - The People's Hospital of Liaoning Province, Shenyang
  - Shaanxi Provincial People's Hospital, Xi'an
  - The Third Affiliated Hospital of Xinjiang Medical University, Xinxiang
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou
  - Yancheng First People's Hospital, Yancheng
  - Yixing People's Hospital, Yixing
  - Yiyang Central Hospital, Yiyang
  - Yueyang Central Hospital, Yueyang
  - Yuncheng Central Hospital, Yuncheng
  - Zibo Municipal Hospital, Zibo